CLINICAL TRIAL: NCT05892679
Title: The Effect of Acupressure on Fatigue, Quality of Life and Comfort in Hemodialysis Patients. Randomized Controlled Study
Brief Title: The Effect of Acupressure in Hemodialysis Patients
Acronym: acupress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, VECİHE DÜZEL GÜNDÜZ, MSN Nurse, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MersinUnv.VDG
Record Dates: First submitted 2023-05-27; First posted 2023-06-07 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Fatigue; Comfort; Quality of Life
Keywords: acupressure; hemodialysis patients; Fatigue; Comfort; Quality of Life
MeSH Terms: conditions — Fatigue | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: The researcher cannot be blinded due to the nature of the research. However, participants will be blinded without knowing whether they are in the study group or the placebo group. Thus, the research will be carried out as a single-blind randomized controlled trial. When the research is completed, the data of the study and control groups (coded as A or B) will be transferred to the computer environment by an independent researcher, and the data will be analyzed by a statistician and the findings will be reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure (Experimental): Acupressure will be formulated according to the standards of the World Health Organization and applied to the determined points in a certain order. Since the reactions of individuals will be different from each other, the stiffness and pressure will be adjusted according to the sensitivity of the individual in order not to cause tissue damage. Pressures will be applied manually by a single practitioner. A total of 8 points with parallel points will be studied, with four points in each lower extremity. There will be a total of 12 minutes of pressure on 8 points, with an average of 90 seconds on each point, and approximately 10-15 seconds of warming and preparatory scrubbing before pressing on the area where the points are located.
  Considering the studies done, a person will be given acupressure three times a week for four weeks.
  Interventions: Other: acupressure
- Control (No Intervention): No intervention will be made to the control group only the data will be collected at the same time as the study group.

INTERVENTIONS:
Other: acupressure — Acupressure will be formulated according to the standards of the World Health Organization and applied to the determined points in a certain order. Since the reactions of individuals will be different from each other, the stiffness and pressure will be adjusted according to the sensitivity of the individual in order not to cause tissue damage. Pressures will be applied manually by a single practitioner. A total of 8 points with parallel points will be studied, with four points in each lower extremity. There will be a total of 12 minutes of pressure on 8 points, with an average of 90 seconds on each point, and approximately 10-15 seconds of warming and preparatory scrubbing before pressing on the area where the points are located.
  Considering the studies done, a person will be given acupressure three times a week for four weeks.
  Arms: Acupressure

SUMMARY:
This randomized controlled study evaluates the effect of acupressure application on fatigue, quality of life and comfort in hemodialysis patients. In our research, it is aimed to reduce fatigue, increase the quality of life and comfort level in hemodialysis patients with acupressure applied.

DETAILED DESCRIPTION:
In the study, 60 hemodialysis patients were randomly assigned to the study and control groups. The study group (n=30) Acupressure is formulated according to the standards of the World Health Organization and in a certain order to the points of Stomach 36 (St 36), Gall Bladder 34 point (GB 34), Spleen 6 point (SP 6) and Kidney 1 point (K 1) will be applied. Consideration will be given to the appropriate pressure intensity and duration. Since the reactions of individuals will be different from each other, the stiffness and pressure will be adjusted according to the sensitivity of the individual in order not to cause tissue damage. Pressures will be applied manually by a single practitioner. Considering the anatomical area where the point is located, the most suitable thumb, index and/or middle finger will be used for application to the relevant point. Successive compressions will be applied at a frequency that does not disturb the patient, does not cause pain, and has a calming effect. Considering the studies done, a person will be given acupressure three times a week for four weeks. No intervention will be made to the control group (n=30). In order to avoid ethical problems both groups will be given an informative training on acupressure and fatigue, increase the quality of life and comfort level in hemodialysis patients at the end of the study. The primary outcome of the study is the effect of acupuncture on fatigue in hemodialysis patients. The secondary result of the study is the effect of acupuncture on quality of life and comfort level in hemodialysis patients.

The results will be collected before the acupressure and in the 4th week of the last intervention.

ELIGIBILITY:
Inclusion Criteria:

* Written and verbal consent was obtained to participate in the study,
* Can read, write, speak and understand Turkish,
* Are older than 18 years,
* Have received HD treatment for at least 6 months,
* Receiving HD treatment 3 times a week,
* Fatigue severity ≥4, using a single-item fatigue index ranging from 0 to 10 points,
* Absence of lower extremity wounds
* Any complementary therapy
* Conscious, fully oriented and cooperative and open to communication,
* No visual, hearing and perception problems,
* Any psychiatric patient

Exclusion Criteria:

* Wound or amputation of lower extremities, rheumatoid arthritis or limb fracture
* Any psychiatric disease,
* Patients with hepatitis B and hepatitis C,
* Using any of the complementary and integrated methods
* Those who receive HD treatment twice a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Fatigue to be evaluated using the Piper Fatigue Scale | Change from before implementation and 4th week of practice
  The total score obtained from the scale varies between 0 and 10 and as the score increases, the fatigue experienced by the individuals increases.

SECONDARY OUTCOMES:
Life Quality to be evaluated using Kidney Disease and Quality of Life Short Form (KDQOL-SF 1.3) | Change from before implementation and 4th week of practice
  Scores on each dimension range from 0 to 100, with higher scores reflecting better health related quality of life.
Comfort to be evaluated using Hemodialysis Comfort Scale | Change from before implementation and 4th week of practice
  The score that can be obtained from the scale varies between 9 and 45. There is an inverse item in the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be used outside of this research.

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT05892679/Prot_SAP_000.pdf
  • Informed Consent Form: INFORMED CONSENT FORM / WORKING GROUP (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT05892679/ICF_001.pdf
  • Informed Consent Form: INFORMED CONSENT FORM / CONTROL GROUP (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT05892679/ICF_002.pdf